CLINICAL TRIAL: NCT00498511
Title: Prospective Evaluation of the Gastrointestinal Tract in Young Men With Iron Deficiency Anemia
Brief Title: Gastrointestinal Evaluation in Young Men With Iron Deficiency Anemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 64/07
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2007-07-13 (Estimated); Status verified 2007-06

CONDITIONS: Anemia, Iron-Deficiency
Keywords: Anemia, Iron-Deficiency; Endoscopy, Gastrointestinal; Male, aged 18 to 40
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Endoscopy, Digestive System; Colonoscopy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: upper gastrointestinal endoscopy, colonoscopy

SUMMARY:
Both upper gastrointestinal endoscopy and colonoscopy are recommended in men and post-menopausal women with iron deficiency anemia. Due to lack of data on the yield of these endoscopies in young men, they are currently investigated as older men. The aim of this study is to evaluate prospectively the prevalence of various gastrointestinal lesions in young men with iron deficiency anemia. Our hypothesis is that the diagnostic yield of colonoscopy in young anemic men without gastrointestinal symptoms is very low, especially if a potential lesion is detected during upper gastrointestinal endoscopy. Therefore, this study will try to identify predicting factors regarding the yield of both endoscopies. Another purpose is to evaluate the outcome of patients with negative endoscopic results, during a follow-up of two years.

ELIGIBILITY:
Inclusion Criteria:

* Men < 40 years old of age with iron deficiency.
* hemoglobin level less than 13 gr/dl documented during the 2 years prior to entering the study with one of the following: 1) iron level less than 45 μg /dl and transferrin saturation less than 10%; 2) ferritin level less than 20 μg/L (both documented during the 4 months prior to entering the study).

Exclusion Criteria:

* Previously diagnosed disease that explain iron deficiency anemia
* Colonoscopy performed during the last 4 years
* Upper gastrointestinal endoscopy performed during the last 2 years

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-08

CONTACTS AND LOCATIONS:
Overall Officials: Alain Nimrod Kimchi, M.D., Principal Investigator — Institute of Gastroenterology and Liver Diseases, Assaf-Harofeh Medical Center, 70300 Zerifin, Israel
Locations (1):
- Institute of Gastroenterology and Liver Diseases, Assaf harofeh Medical Center, Ẕerifin, Israel